CLINICAL TRIAL: NCT00411099
Title: An 8-week, Randomized, Double-blind, Fixed Dosage, Placebo-controlled, Parallel-group, Multi-center Study of the Efficacy, Safety and Tolerability of Agomelatine 25 mg and 50 mg in the Treatment of Major Depressive Disorder (MDD) Followed by a 52-week, Open-label Extension (CAGO178A2301E)
Brief Title: Efficacy, Safety and Tolerability of Agomelatine in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAGO178A2301
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
Keywords: agomelatine, major depressive disorder, MDD, depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — agomelatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: agomelatine
- 2 (Experimental)
  Interventions: Drug: agomelatine
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: agomelatine
  Arms: 1; 2
Drug: placebo
  Arms: 3

SUMMARY:
This study will assess efficacy, safety and tolerability of agomelatine (AGO178) 25 mg and 50 mg in patients with Major Depressive Disorder (MDD). This study includes an 8-week double-blind phase and a 52-week open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder, single or recurrent episode, according to DSM-IV criteria
* HAM-D17 total score > or = 22 at Screening and Baseline
* CGI-Severity score > or = 4 at Screening and Baseline
* Only patients who complete the core protocol are eligible to participate in the Open-Label Extension Phase

Exclusion Criteria:

* History of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder, or obsessive compulsive disorder
* Any current Axis I disorder other than major depressive disorder which is the focus of treatment
* Substance or alcohol abuse in the last 30 days, dependence in the last 6 months
* Concomitant psychotropic medication, including herbal preparations and melatonin
* Psychotherapy of any type
* Female patients of childbearing potential who are not using effective contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the change from Baseline to Week 8 on the total score of the clinician rated 17-Item Hamilton Depression Rating Scale (HAM-D17) | 8 weeks

SECONDARY OUTCOMES:
To evaluate the proportion of patients who demonstrate clinical improvement at Week 8, where improvement is defined by a score of 1 or 2 on the CGI-I scale | 8 weeks
To evaluate the proportion of patients who achieve remission at Week 8, where remission is defined by a total score of < or =7 on the HAM-D17 | 8 weeks
To evaluate efficacy with respect to the proportion of patients who demonstrate clinical response, where response is defined by a reduction of at least 50% in the baseline HAM-D17 at week 8 | 8 weeks
To evaluate the change from baseline to week 8 on the subscale scores (Maier, anxiety, retardation and sleep) of the clinician-rated HAM-D17 | 8 weeks
To evaluate subjective sleep (onset and quality), as measured by the scores on the Leeds Sleep Evaluation Questionnaire (LSEQ) at week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (41):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Cerritos, California
  - Novartis Investigative Site, El Centro, California
  - Novartis Investigative Site, Garden Grove, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, Lafayette, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Temecula, California
  - Novartis Investigative Site, Cromwell, Connecticut
  - Novartis Investigative Site, Hamden, Connecticut
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Maitland, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Salisbury, Maryland
  - Novartis Investigative Site, Pittsfield, Massachusetts
  - Novartis Investigative Site, Farmington Hills, Michigan
  - Novartis Investigative Site, Rochester Hills, Michigan
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - Novartis Investigative Site, Princeton, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Beachwood, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Bennington, Vermont
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Bothell, Washington
- Puerto Rico (2):
  - Novartis Investigative Site, Bayamón
  - Novartis Investigative Site, Rio Piedras

REFERENCES:
- See also: Results for CAGO178A2301 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2625